CLINICAL TRIAL: NCT04870710
Title: Improving Visual Hallucinations by Targeting the Visual Cortex With Electrical Stimulation: A Feasibility Study
Brief Title: Feasibility Electrical Stimulation Study for Visual Hallucinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Paulo Lizano, Assistant Professor of Psychiatry, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2019P001016; UL1TR002541 (NIH)
Record Dates: First submitted 2021-04-16; First posted 2021-05-03 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- cathodal transcranial direct current stimulation (tDCS) (Experimental): Two, twenty minute sessions of cathodal tDCS to the bilateral extrastriate visual cortex for 5 days (10 total sessions).
  Interventions: Device: transcranial electrical stimulation
- Anodal transcranial alternating current stimulation (tACS) (Experimental): Two, twenty minute sessions of anodal tACS delta phase aligned for 5 days (10 total sessions).
  Interventions: Device: transcranial electrical stimulation

INTERVENTIONS:
Device: transcranial electrical stimulation — Electrical stimulation to the extrastriate visual cortex.

SUMMARY:
The visual system has increasingly been recognized as an important site of injury in patients with schizophrenia and other psychoses. Visual system alterations manifest as visual perceptual aberrations, deficits in visual processing, and visual hallucinations. These visual symptoms are associated with worse symptoms, poorer outcome and resistance to treatment. A recent study using brain lesion mapping of visual hallucinations and identified a causal location in the part of the brain that processes visual information (visual cortex). The association between visual cortex activation and visual hallucinations suggests that this region could be targeted using noninvasive brain stimulation. Two case studies have found that brain stimulation to the visual cortex improved visual hallucinations in treatment resistant patients with psychosis. While promising it is unclear whether these symptom reductions resulted from activity changes in the visual cortex or not. Here we aim to answer the question whether noninvasive brain stimulation when optimally targeted to the visual cortex can improve brain activity, visual processing and visual hallucinations. The knowledge gained from this study will contribute to the field of vision by providing a marker for clinical response and by personalizing treatment for patients with psychosis suffering from visual symptoms. This grant will allow us to set the foundation for a larger more targeted study utilizing noninvasive brain stimulation to improve visual symptoms in patients with psychosis.

DETAILED DESCRIPTION:
The visual system has increasingly been recognized as an important site of pathology in patients with schizophrenia and other psychoses. Visual system impairments manifest as visual perceptual aberrations, deficits in visual processing tasks, and visual hallucinations (VH). In psychosis spectrum disorders, increased visual aberrations are strongly correlated with worse hallucinations and delusions. It is also recognized that poorer performance on visual spatial working memory, visual integration, and velocity discrimination tasks are associated with greater negative symptoms (a major contributor to disability). VH are common in psychotic disorders (30-70% prevalence) and can be refractory to existing treatments. VH have been understudied in psychosis with much of the literature focusing on auditory hallucinations. Despite the neuroscientific and clinical significance of VH, the brain regions responsible are less clear.

Functional neuroimaging studies have identified neural correlates of VH across multiple brain regions (lingual, fusiform, cuneus, lateral geniculate nucleus, and occipital cortex) and support hypotheses that increased visual cortex activity and sensory cortex over-stimulation generate VH. However, whether these neuroimaging findings represented a cause, consequence or incidental correlate of VH was unclear until recently. Using a newly validated technique termed lesion network mapping, researchers demonstrated that focal brain lesions having a causal role in the development of VH can occur in different brain locations, both inside and outside sensory pathways, and that these lesions are functionally connected to the lateral geniculate nucleus, a major relay center for the visual pathway. They also found that 98% of the subcortical and cortical lesions were connected to the exact same location in the extrastriate visual cortex. Therefore, the association between extrastriate visual cortex activation and VH would suggest this region may be optimal for modulation via brain stimulation.

One method by which cortical excitability can be altered is through the use of transcranial electrical stimulation (tES), a non-invasive brain stimulation technique. High definition tES (HD-tES) is a refined version of tES with improved spatial precision of cortical stimulation. This involves the application of a weak electrical current (1-2 mA) delivered to the brain via scalp electrodes. The effects of tES modulate cortical excitability where anodal stimulation tends to increase (i.e. the resting potential becomes less negative) and cathodal stimulation tends to decrease the underlying membrane potential (i.e. the resting potential becomes more negative) (14,15). Studies have shown that tES can modulate visual cortical function in a polarity-dependent manner, where anodal stimulation can increase and cathodal stimulation can decrease the amplitude of the N70 component from the visual-evoked potential. While tES is a promising adjunctive treatment of auditory hallucinations and negative symptoms in schizophrenia, less is known about its role in treating VH. To date, two cases have been described where cathodal tES (i.e., outward current flow) over the occipital area was applied to patients experiencing treatment refractory VH, and this resulted in symptomatic improvement. Taken together, the recent lesion network mapping identifying the extrastriate visual cortex as a major source of VH in schizophrenia combined with these two single-patient case studies suggest that it may be possible to alleviate VH by designing a tES protocol that targets the extrastriate visual cortex bilaterally. Technological advances in noninvasive neuromodulation and electrical field modeling further allow us to create a tES protocol specifically guided by the results of lesion network mapping studies (i.e., using the exact Montreal Neurological Institute coordinates) with high spatial resolution (i.e., using HD-tES).

ELIGIBILITY:
Inclusion Criteria:

* meet diagnostic criteria for schizophrenia, schizoaffective disorder, or psychotic bipolar disorder as verified by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV TR) and consensus clinical diagnosis;
* had no changes to relevant anti-psychotic medications for a period of 1 month prior to participation;
* had a sufficient level of English to allow participation.

Exclusion Criteria:

* pregnant or breastfeeding women;
* Intelligence quotient <60
* any major medical or neurologic
* diagnosis of substance abuse positive urine drug screen
* history of moderate-to-severe visual impairment secondary to glaucoma, cataract or macular degeneration
* serious medical illness or instability requiring hospitalization within the next year
* relevant skin allergies; metallic or electronic implants (e.g. pacemakers, brain stimulators).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Lizano, MD,PhD, Principal Investigator — Staff Physician/Scientist
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raymond N, Reinhart RMG, Trotti R, Parker D, Grover S, Turkozer B, Sabatinelli D, Hegde R, Bannai D, Gandu S, Clementz B, Keshavan M, Lizano P. Efficacy and Tolerability of Lesion Network Guided Transcranial Electrical Stimulation in Outpatients with Psychosis Spectrum Illness: A Nonrandomized Controlled Trial. medRxiv [Preprint]. 2023 Apr 3:2023.03.31.23287980. doi: 10.1101/2023.03.31.23287980. PMID 37066217

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment efforts ended prior to the end of the trial (Jan 2, 2022) resulting with 6 individuals who met criteria for schizophrenia, schizoaffective or bipolar disorder entering the study. Recruitment efforts were done through utilizing past research repositories and individuals were contacted through email or phone. Interested individuals were then phone screened for additional study criteria including safety to receive transcranial electrical stimulation (tES) and current symptoms.
Pre-assignment Details: Participants were first consented and met with a trained medical professor review any medical changes or relevant changes to diagnosis to ensure safe measures for tES treatment. Individuals who were recruited were then requested to completed a clinical assignment as well as baseline measurements for EEG and behavioral tasks before receiving any tES treatment.
Groups:
- Transcranial Electrical Stimulation (tES): Two, twenty minute sessions of cathodal cathodal transcranial direct current stimulation (tDCS) to the bilateral extrastriate visual cortex for 5 days (10 total sessions). After which individuals entered the transcranial alternating current stimulation (tACS) arm of the study which followed the same treatment parameters as the tDCS arm.
  transcranial electrical stimulation: Electrical stimulation to the extrastriate visual cortex.
Period: Overall Study
Arm/Group | Transcranial Electrical Stimulation (tES)
Started | 6
Transcranial Direct Current Stimulation (tDCS) Baseline Assessment | 6
Transcranial Direct Current Stimulation (tDCS) Five Day Follow-up Assessment | 6
Transcranial Direct Current Stimulation (tDCS) 1 Month Follow-up Assessment | 5
Transcranial Alternating Current Stimulation (tACS) Baseline Assessment | 4
Transcranial Alternating Current Stimulation (tACS) 5 Day Follow up Assessment | 4
Transcranial Alternating Current Stimulation (tACS) 1 Month Follow up Assessment | 3
Completed | 3
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: The total number of participates recruited was 6 individuals. However, we utilized a cross-over design with 6 individuals completing the cathodal tDCS condition (baseline and day 5) and 4 individuals completing the tACS condition (baseline and day 5) .
Groups:
- Transcranial Electrical Stimualtion: After participants performed a clinical assignment, EEG and behavioral tasks they were entered into the treatment phase of the study. Individuals first received two, twenty minute sessions of cathodal tDCS to the bilateral extrastriate visual cortex for 5 days (10 total sessions). After which, and additional clinical assignment, EEG and behavioral task battery were performed on day 5. Participants were then asked to come back in a month for an additional follow up visit that consisted of a clinical assignment, EEG and behavioral task battery. Participants were then scheduled to entered the 2hz tACS condition after they completed a minimum 2 week washout period. individuals were allocated to receive two, twenty minute sessions of 2hz tACS to the bilateral extrastriate visual cortex for 5 days (10 total sessions). At day 5, another clinical assignment, EEG and behavioral task battery was preformed. Participants were then asked to come back after 1month to receive an additional follow up visit.
Arm/Group | Transcranial Electrical Stimualtion
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.67 (2.58)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 2
  Female | 3
  Transgender | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Steady State Visual Evoked Potential (ssVEP)
Description: Measuring the average evoked response potential amplitude change for P100 at Baseline, 5 day and 1 month visits. ssVEP was utilized to measure changes in electrical biomarkers of the early visual response. Stimuli consisted of 50 trials of a black and white square oscillating at 18.75 Hz in the subject's central, bilateral, left, or right visual field for 2000 ms (200 total trials pseudorandomly interleaved) with inter-trial intervals of 2.5 seconds.
Time Frame: Measured at day 5 compared to day 0
Measure: Median (Inter-Quartile Range); unit: microvolts
Arm/Group | Cathodal Transcranial Direct Current Stimulation (tDCS) | Anodal Transcranial Alternating Current Stimulation (tACS)
Number analyzed (Participants) | 6 | 4
microvolts
  Baseline | 1.725 [0.910 to 3.035] | 1.160 [0.480 to 2.933]
  Day 5 | 1.180 [0.503 to 2.053] | 1.005 [0.483 to 3.238]
Statistical Analysis 1: Comparison: Cathodal Transcranial Direct Current Stimulation (tDCS) vs Anodal Transcranial Alternating Current Stimulation (tACS); Test type: Superiority; p = 0.10, Friedman; Median Difference (Net) = 0.10; Non-parametric tests were used consisting of Friedman and Durbin Conover tests

2. Primary Outcome: Steady State Visual Evoked Potential (ssVEP)
Description: as for outcome 1
Time Frame: Measured at day 30 compared to day 0 and day 5
Measure: Median (Inter-Quartile Range); unit: microvolts
Arm/Group | Cathodal Transcranial Direct Current Stimulation (tDCS) | Anodal Transcranial Alternating Current Stimulation (tACS)
Number analyzed (Participants) | 6 | 4
microvolts
  Baseline | 1.725 [0.910 to 3.035] | 1.160 [0.480 to 2.933]
  5 day | 1.180 [0.503 to 2.053] | 1.005 [0.483 to 3.238]
  1 Month | 1.160 [0.218 to 2.860] | 2.560 [1.035 to 4.412]

3. Primary Outcome: Positive and Negative Syndrome Scale (PANSS)
Description: Measuring total psychosis symptoms score. PANSS is a clinician administered instrument which has 30 items measuring a range of symptoms which are rated on a 7-point scale (1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, and 7=extreme). A total score ranges from 30-210 with higher scores indicate worsen symptoms. Subscales include, general, negative and positive symptom categories with higher scores indicate worsen symptoms. The range for the positive and negative Scales is 7-49, and the range for the general Psychopathology Scale is 16-112.
Time Frame: Measured at day 5 compared to day 0
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cathodal Transcranial Direct Current Stimulation (tDCS) | Anodal Transcranial Alternating Current Stimulation (tACS)
Number analyzed (Participants) | 6 | 4
score on a scale
  Baseline | 49.50 [43.50 to 59.25] | 59.50 [54.50 to 67.50]
  5 Day | 44.00 [40.50 to 49.75] | 56.50 [50.50 to 64.75]

4. Primary Outcome: Positive and Negative Syndrome Scale (PANSS)
Description: as for outcome 3
Time Frame: Measured at day 30 compared to day 0 and day 5
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Cathodal Transcranial Direct Current Stimulation (tDCS) | Anodal Transcranial Alternating Current Stimulation (tACS)
Number analyzed (Participants) | 6 | 4
units on a scale
  Baseline | 49.50 [43.50 to 59.25] | 59.50 [54.50 to 67.50]
  Day 5 | 44.00 [40.50 to 49.75] | 56.50 [50.50 to 64.75]
  1 Month | 50.00 [48.25 to 54.75] | 47.50 [43.75 to 52.00]

5. Primary Outcome: Biological Motion
Description: Measuring the percent correct of detected motion. Biological motion perception was assessed using point-light animations (12 dots on the head and major joints of the body) walking either rightward or leftward. The target animation was embedded in a number of random-moving noise dots (24, 48, or 72) to manipulate the difficulty level of the task. Participants were asked to indicate the direction that the animation was walking towards. The task lasted for about 4 minutes.
Time Frame: Measured at day 5 compared to day 0
Measure: Median (Inter-Quartile Range); unit: percentage of correct responses
Arm/Group | Cathodal Transcranial Direct Current Stimulation (tDCS) | Anodal Transcranial Alternating Current Stimulation (tACS)
Number analyzed (Participants) | 6 | 4
percentage of correct responses
  Baseline | 63.33 [57.08 to 70.83] | 60.00 [52.50 to 69.17]
  5 Day | 68.33 [58.33 to 77.08] | 71.67 [63.33 to 79.17]

6. Primary Outcome: Biological Motion
Description: as for outcome 5
Time Frame: Measured at day 30 compared to day 0 and day 5
Measure: Median (Inter-Quartile Range); unit: percentage of correct responses
Arm/Group | Cathodal Transcranial Direct Current Stimulation (tDCS) | Anodal Transcranial Alternating Current Stimulation (tACS)
Number analyzed (Participants) | 6 | 4
percentage of correct responses
  Baseline | 63.33 [57.08 to 70.83] | 60.00 [52.50 to 69.17]
  5 Day | 68.33 [58.33 to 77.08] | 71.67 [63.33 to 79.17]
  1 Month | 69.17 [62.50 to 78.33] | 60.00 [59.17 to 74.17]

7. Secondary Outcome: International Affective Picture System (IAPS) Task
Description: Emotional evoked related potential (ERP) measures were obtained using the IAPS, which consists of unpleasant, pleasant, and neutral scene stimuli. Scenes consisted of human threat, animal threat, erotica, romantic couples, people, families, and landscapes. During each experimental session, participants viewed each scene three times. Images were presented for 1000 ms and then followed by 3.5 s of a black screen with a small red dot as a fixation point.
Time Frame: Measured at day 5 compared to day 0
Population: 1 individual in our sample pool did not feel comfortable completing the task, leaving us with 5 individuals in the tDCS condition for analysis. Too few individuals in the tACS completed the task for effective analysis and data was deemed poor quality or insufficient to process.
Measure: Median (Inter-Quartile Range); unit: microvolts
Arm/Group | Cathodal Transcranial Direct Current Stimulation (tDCS) | Anodal Transcranial Alternating Current Stimulation (tACS)
Number analyzed (Participants) | 5 | 0
microvolts
  Baseline | 6.525 [6.348 to 6.787] |
  5 Day | 5.751 [5.139 to 5.856] |

8. Secondary Outcome: International Affective Picture System (IAPS) Task
Description: as for outcome 7
Time Frame: Measured at day 30 compared to day 0 and day 5
Population: 1 individual in our sample pool did not feel comfortable completing the task, leaving us with 5 individuals in the tDCS condition for analysis. Too few individuals in the tACS completed the task for effective analysis and data that was collected was insufficient quality to process through software.
Measure: Median (Inter-Quartile Range); unit: microvolts
Arm/Group | Cathodal Transcranial Direct Current Stimulation (tDCS) | Anodal Transcranial Alternating Current Stimulation (tACS)
Number analyzed (Participants) | 5 | 0
microvolts
  Baseline | 6.525 [6.348 to 6.787] |
  5 Day | 5.751 [5.139 to 5.856] |
  1 Month | 3.25 [3.247 to 4.348] |

9. Secondary Outcome: Velocity Discrimination
Description: Velocity discrimination performance was determined using constant stimuli method. Participants asked to indicate the faster of the two gradients (drifting Gabor patches) presented sequentially for 300 ms with an inter-stimulus interval of 500ms 51.There were 9 velocity difference levels to modulate the difficulty of the task. 15 trials were presented at each difficulty level. Velocity discrimination thresholds, which corresponds to an accuracy level equivalent to 75% correct for each subject, calculated as an indicator of performance. This task session lasted for about 5 minutes.
Time Frame: Measured at day 5 compared to day 0
Population: Too few individuals met threshold requirements related to task to perform analysis for Velocity Discrimination due to insufficient data/poor quality or participant drop out.
Measure: Median (Inter-Quartile Range); unit: percentage of total correct
Arm/Group | Cathodal Transcranial Direct Current Stimulation (tDCS) | Anodal Transcranial Alternating Current Stimulation (tACS)
Number analyzed (Participants) | 5 | 3
percentage of total correct
  Baseline | 0.181 [0.123 to 0.205] | 0.2020 [0.1510 to 0.2160]
  5 Day Follow up | 0.188 [0.168 to 0.218] | 0.1600 [0.0875 to 0.1700]

10. Secondary Outcome: Velocity Discrimination
Description: as for outcome 9
Time Frame: Measured at day 30 compared to day 0 and day 5
Population: Too few individuals met threshold requirements related to task to perform analysis for Velocity Discrimination. This was due to insufficient data/poor quality or participant drop out.
Measure: Median (Inter-Quartile Range); unit: percentage of total correct
Arm/Group | Cathodal Transcranial Direct Current Stimulation (tDCS) | Anodal Transcranial Alternating Current Stimulation (tACS)
Number analyzed (Participants) | 5 | 3
percentage of total correct
  Baseline | 0.181 [0.123 to 0.205] | 0.2020 [0.1510 to 0.2160]
  5 Day | 0.188 [0.168 to 0.218] | 0.1600 [0.0875 to 0.1700]
  1 Month | 0.188 [0.167 to 0.202] | 0.17 [0.17 to 0.17]

11. Secondary Outcome: Visual Spatial Working Memory
Description: To assess visuospatial working memory participants were asked to identify and remember the location of the odd shape out of three shapes. The procedure was repeated with three new shapes following an interval. Participants were asked to respond by indicating where the odd shapes appeared, in the correct order of appearance. Two correct trials on each level led to progression to the next level where the item load was increased by one. The session was terminated when two trials on the same level were incorrect. The final score was calculated based on the performance on the highest level achieved (10 max) where at least one trial was passed. A higher score means better visual spatial memory capability (0-10) and the highest difficulty level achieved. This task lasted for 3-5 minutes.
Time Frame: Measured at day 5 compared to day 0
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cathodal Transcranial Direct Current Stimulation (tDCS) | Anodal Transcranial Alternating Current Stimulation (tACS)
Number analyzed (Participants) | 6 | 4
score on a scale
  Baseline | 5.925 [4.763 to 6.300] | 5.000 [4.775 to 5.125]
  5 Day | 5.250 [4.612 to 5.700] | 4.700 [4.275 to 5.050]

12. Secondary Outcome: Visual Spatial Working Memory
Description: as for outcome 11
Time Frame: Measured at day 30 compared to day 0 and day 5
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cathodal Transcranial Direct Current Stimulation (tDCS) | Anodal Transcranial Alternating Current Stimulation (tACS)
Number analyzed (Participants) | 6 | 4
score on a scale
  Baseline | 5.925 [4.763 to 6.300] | 5.000 [4.775 to 5.125]
  Day 5 | 5.250 [4.612 to 5.700] | 4.700 [4.275 to 5.050]
  1 Month | 6.475 [5.612 to 7.300] | 5.250 [4.900 to 5.325]

13. Secondary Outcome: Global Assessment of Function (GAF)
Description: Measuring global functioning derived from patients symptoms, relationships and functioning in life. The higher the score, the better individual handles daily activities and lower symptoms experienced.
  91-100 No symptoms. Superior functioning in a wide range of activities. 81-90 Absent or minimal symptoms, good functioning in all areas. 71-80 Symptoms are transient and expectable reactions to psychosocial stressors.
  61-70 Some mild symptoms or some difficulty in functioning. 51-60 Moderate symptoms or moderate difficulty in functioning. 41-50 Serious symptoms or any serious impairment in functioning 31-40 Some impairment or major impairment in several areas, such as work or school, family relations, judgment, thinking, or mood.
  21-30 Behavior is considerably influenced by delusions or hallucinations or serious impairment 11-20 Some danger of hurting self or others. 1-10 Persistent danger of severely hurting self or others. 0 Inadequate information
Time Frame: Measured at day 5 compared to day 0
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cathodal Transcranial Direct Current Stimulation (tDCS) | Anodal Transcranial Alternating Current Stimulation (tACS)
Number analyzed (Participants) | 6 | 4
score on a scale
  Baseline | 70.00 [62.00 to 78.75] | 65.00 [60.00 to 66.25]
  5 Day | 68.50 [61.25 to 78.75] | 65.00 [61.75 to 66.25]

14. Secondary Outcome: Global Assessment of Function (GAF)
Description: as for outcome 13
Time Frame: Measured at day 30 compared to day 0 and day 5
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cathodal Transcranial Direct Current Stimulation (tDCS) | Anodal Transcranial Alternating Current Stimulation (tACS)
Number analyzed (Participants) | 6 | 4
score on a scale
  Baseline | 70.00 [62.00 to 78.75] | 65.00 [60.00 to 66.25]
  5 Day | 68.50 [61.25 to 78.75] | 65.00 [61.75 to 66.25]
  1 Month | 63.00 [53.50 to 65.00] | 68.00 [65.75 to 72.50]

15. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Measuring total depression scores, The Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire which psychiatrists or trained mental health providers use to measure the severity of depressive episodes and or symptoms in patients with mood disorders. A higher score indicates worsen depression.
  The questionnaire includes questions on ten symptoms:Apparent sadness, Reported sadness, Inner tension, Reduced sleep, Reduced appetite, Concentration difficulties, Lassitude, Inability to feel, Pessimistic thoughts, Suicidal thoughts.
  Total used from scale indicates:
  0 to 6: normal/symptom absent 7 to 19: mild depression 20 to 34: moderate depression 35 to 60: severe depression
Time Frame: Measured at day 5 compared to day 0
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cathodal Transcranial Direct Current Stimulation (tDCS) | Anodal Transcranial Alternating Current Stimulation (tACS)
Number analyzed (Participants) | 6 | 4
score on a scale
  Baseline | 6.00 [4.25 to 15.25] | 5.50 [3.75 to 10.00]
  5 Day | 3.50 [3.00 to 5.50] | 4.00 [2.25 to 8.00]

16. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: as for outcome 15
Time Frame: Measured at day 30 compared to day 0 and day 5
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Cathodal Transcranial Direct Current Stimulation (tDCS) | Anodal Transcranial Alternating Current Stimulation (tACS)
Number analyzed (Participants) | 6 | 4
units on a scale
  Baseline | 6.00 [4.25 to 15.25] | 5.50 [3.75 to 10.00]
  Day 5 | 3.50 [3.00 to 5.50] | 4.00 [2.25 to 8.00]
  1 Month | 6.00 [2.00 to 7.75] | 2.50 [0.00 to 5.50]

ADVERSE EVENTS:
Time Frame: Data related to adverse events were collected up to study completion or at each assessment time point (baseline, day 5 and 1month)
Description: Participants performed clinical assessments at baseline, 5 day and 1 month which tracked symptoms of psychosis, depression and others through standard and valid clinical assessments tools by trained providers. Additionally, study team members utilized a sensation form related to tES treatment. Each participant was required to fill out a sensation questionnaire after each tES session.
Groups:
- 2hz Transcranial Alternating Current Stimulation (tACS): Two, twenty minute sessions of 2hz tACS delta for 5 days (10 total sessions).
  transcranial electrical stimulation: Electrical stimulation to the extrastriate visual cortex.
Arm/Group | Cathodal Transcranial Direct Current Stimulation (tDCS) | 2hz Transcranial Alternating Current Stimulation (tACS)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 0/6 | 0/4

LIMITATIONS AND CAVEATS:
Our main analysis included individuals with imputed values for follow up visits (1 individual for 1 month tDCS; 1 individual for 1 month tACS).

Due to corona virus related regulations our recruitment was hindered and resulted in a small sample size.

Individuals were recruited from a single site. Recruited individuals were mainly stable during their baseline clinical assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-01-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT04870710/Prot_001.pdf